CLINICAL TRIAL: NCT01724047
Title: Autism Intervention Research Network for Behavioral Health (AIR-B II): Network Activity A: Conduct Research on Evidence-Based Practices.
Brief Title: Autism Intervention Research Network for Behavioral Health (AIR-B II): Deployment Into Elementary Schools
Acronym: AIR-B II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Health Resources and Services Administration (HRSA) (U.S. Federal Agency)
Collaborators: University of Rochester (Other); University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Connie Kasari, Ph.D., Professor, University of California, Los Angeles
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 12-001120
Record Dates: First submitted 2012-11-05; First posted 2012-11-09 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Autism
Keywords: Autism; School Based Intervention
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Playground Intervention (Experimental): Schools will be randomized to one of two conditions. The conditions are: 1) Immediate treatment, where the training will begin immediately after baseline measures are completed 2) Waitlist treatment, where the training will begin the following school year. The initial delivery will occur for 30 minutes three times for a period of two to three weeks, then 30 minutes two times for a period of two weeks, then 30 minutes once a week for up to 16 sessions, within a period of 3 months, then a 30 minute follow up will occur 3 months later. A systematic fading of intervention using performance feedback, coaching, and consultation. Outcome measures will be administered at entry, end of treatment, and 3-month follow-up. Entry diagnostic, exit and follow up assessments will last 1.5- 2 hours and participants will be assessed after school or in their homes.
  Interventions: Behavioral: Playground Intervention
- STAT Intervention (Experimental): Classrooms will be randomized to one of two conditions. The conditions are: 1) Immediate treatment, where the training will begin immediately after baseline measures are completed. 2) Waitlist treatment, where the training will begin the following school year. The intervention will be over a period of 6 weeks, with baseline, treatment, and a follow up visit totaling 18 weeks at the school site. Each visit is approximately 30 minutes. A systematic fading of intervention using performance feedback, coaching, and consultation. Outcome measures will be administered at entry, end of treatment. Entry diagnostic, exit and follow up assessments will last 1.5- 2 hours and participants will be assessed after school or in their homes.
  Interventions: Behavioral: STAT Intervention
- Playground Waitlist Control (No Intervention): Waitlist Control
- STAT Waitlist Control (No Intervention): Waitlist Control

INTERVENTIONS:
Behavioral: Playground Intervention — Intervention is designed for children diagnosed with an autism spectrum disorder (ASD) included in a regular education k through fifth grade classroom for at least 50% of the school day. Schools will be randomized to one of two conditions. The conditions are: 1) Immediate treatment, where the training will begin immediately after baseline measures are completed. 2) Waitlist treatment, where the training will begin the following school year. This study will take place at school. All intervention activities will be conducted during recess or lunch where children with autism may have the most difficulty interacting with peers. A total of 14-16 intervention sessions will be held with the child with autism, school personnel, and the child's classmates. The intervention will last approximately 3 months with a 3-month follow-up.
  Arms: Playground Intervention
Behavioral: STAT Intervention — This study will track the behavioral progress of children whose teachers receive training in these instructional methods. This study also will examine the ability and willingness of teachers to use these methods as they were designed. The study will last approximately 18 weeks (6 weeks of intervention, and a 3 month follow up visit). This study will take place at school. Classrooms will be randomized to one of two conditions. The conditions are: 1) Immediate treatment, where the training will begin immediately after baseline measures are completed. 2) Waitlist treatment, where the training will begin the following school year. All intervention activities will be conducted with a teacher during the school day but not during instructional time. Study staff will visit the school on a weekly basis to train your child's teacher on evidence-based strategies for teaching children with autism.
  Arms: STAT Intervention

SUMMARY:
The primary goal of this study is to identify efficacious and cost effective intervention strategies that can improve academic and psychological outcomes for children with ASD, and can be feasibly be implemented at fidelity by school personnel in under served elementary schools. Two simultaneous interventions will occur.

In intervention 1, students with ASD in inclusion classrooms will be randomized to the Playground Intervention or a waitlist control group. In the Playground Intervention, UCLA/ROC/UPENN staff will work with school personals (teachers, paraprofessionals) to increase peer engagement on the yard.

In intervention 2, students in special day classes will be randomized to the 'Schedule Tools Activities Transitions' Intervention (STAT) or wait-list control. In the STAT Intervention, UCLA/ROC/UPENN staff will work with teachers to implement behavioral strategies in the classrooms.

In both interventions, the conditions are: 1) Immediate treatment, where the training will begin immediately after baseline measures are completed. 2) Wait-list treatment, where the training will begin the follow school year.

ELIGIBILITY:
Inclusion Criteria:

1. Child: Child has to meet the following criteria: 1) Child's primary classroom teacher has consented to participate, 2) Child meets ADOS research criteria for autism spectrum disorder, 3) Child is between 5-11 years old, 4) Child's parents consented to have child participate, and 5) Child is placed in inclusion classroom or self-contained special education classroom for a minimum of 50% of the school day.
2. Adult: School teachers and paraprofessionals working with children with ASD.

Exclusion Criteria:

1. Child: Participants will be excluded from the study if child has co-morbid disorders such as cerebral palsy, Fragile X, Down syndrome. Child has profound vision or hearing lose.
2. Adult: Participants will be excluded from the study if the adult is not a teacher, administrator, teaching assistant, yard attendant, related services provider, or a paraprofessional.

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2012-11; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Playground Intervention: Playground Peer Engagement | Change from baseline to exit (12 weeks later) in the POPE
  Playground Intervention: Peer Observation of Playground Engagement (POPE) measure. Peer interactions on the playground will be coded using an interval-observation schedule of every 40 seconds (with 20 second coding intervals). Interactive levels or states will be noted along with the presence or absence of discrete interactive behaviors during each coding interval.
Playground Intervention: Playground Peer Engagement | Change from exit to follow up (3 months later) in the POPE
  Playground Intervention: Peer Observation of Playground Engagement (POPE) measure. Peer interactions on the playground will be coded using an interval-observation schedule of every 40 seconds (with 20 second coding intervals). Interactive levels or states will be noted along with the presence or absence of discrete interactive behaviors during each coding interval.
Playground Intervention: Social Network Salience | Change from baseline to exit (12 weeks later) in Playground Intervention Social Network
  Playground Intervention: Social Network measure. Based on the Cairns' (1994) method, participants will be asked to list all the names of children in their class who hang out together; this free-recall method is used rather than asking respondents to place each peer's name in a group, because the relative strength of students' tendency to recall classmates is an important indicator of the peers' prominence in the social structure.
Playground Intervention: Social Network Salience | Change from exit to follow up (3 months later) in Playground Intervention Social Network
  Playground Intervention: Social Network Measure. Based on the Cairns' (1994) method, participants will be asked to list all the names of children in their class who hang out together; this free-recall method is used rather than asking respondents to place each peer's name in a group, because the relative strength of students' tendency to recall classmates is an important indicator of the peers' prominence in the social structure.
STAT Intervention: Teacher Behaviors and Student's Engagement in the Classrooms | Change from Baseline to Exit (6 weeks later) in STAT Intervention: Classroom Observational Measure
  STAT Intervention: The Classroom Observational Measure is an adaptive observational measure designed to capture teacher behaviors and student behaviors in the classroom that includes teacher's praises, behavioral control and student's on/off task behaviors.
STAT Intervention: Teacher Behaviors and Student's Engagement in the Classrooms | Change from Exit to Follow Up (3 months later) in STAT Intervention: Classroom Observational Measure
  STAT Intervention: The Classroom Observational Measure is an adaptive observational measure designed to capture teacher behaviors and student behaviors in the classroom that includes teacher's praises, behavioral control and student's on/off task behaviors.

SECONDARY OUTCOMES:
Playground Intervention: Teachers Ratings of Intervention Implementation | Exit (12 weeks from Baseline)
  Playground Intervention Teacher Implementation Climate Measure. Climate for Implementation Measure is a 17-item questionnaire to measure the climate of each classroom. The survey asks teachers and aides to rate their perception of program quality and ease of use, and global perceptions of staff climate.
Playground Intervention: Teacher's Perceptions of Intervention | Change from baseline to exit (12 weeks later) in Playground Intervention Teacher Perception of Intervention
  The teacher perception of social skill (TPSS) is a 26-item questionnaire that uses a 3-point Likert scale to rate 12 items regarding teachers' perceptions of participants' social skills (1 = never, 2 = sometimes and 3 = very often). The social skills domain describes the child's strengths, such as adaptability to the school classroom and environment, quality of interactions with peers, and popularity or likeability among peers (Sorongon, Kim, & Zill, 2000).
STAT Intervention: Teacher Nominated Target Behaviors | Change from baseline to exit (6 weeks later) in STAT Intervention: Teacher Nominated Target Behaviors
  Teacher report of student's behavioral problems in the classroom.
STAT Intervention: Teacher Nominated Target Behaviors | Change from Exit to Follow Up (3 months later) in STAT Intervention Classroom Observational Measure
  STAT Intervention: Classroom Observational Measure is an adaptive observational measure designed to capture teacher behaviors and student behaviors in the classroom.
Playground Intervention Teacher's Perceptions of Intervention | Change from exit to follow up (3 months later) in Playground Intervention Teacher Perception of Intervention
  The teacher perception of social skill (TPSS) is a 26-item questionnaire that uses a 3-point Likert scale to rate 12 items regarding teachers' perceptions of participants' social skills (1 = never, 2 = sometimes and 3 = very often). The social skills domain describes the child's strengths, such as adaptability to the school classroom and environment, quality of interactions with peers, and popularity or likeability among peers (Sorongon, Kim, & Zill, 2000).
STAT Intervention: Teacher Nominated Target Behaviors | Change from exit to follow up (3 months later) in STAT Intervention: Teacher Nominated Target Behaviors
  Teacher report of student's behavioral problems in the classroom.
Playground Intervention: Coach Ratings of Aide Implementation | Change from Baseline to Exit (12 weeks later) in Playground Intervention Coach Rated Aide Fidelity
  Playground Intervention-Coach Rated Aide Fidelity. Fidelity forms will measure implementation mastery of interventionists and school personnel. This is to ensure that interventionists are teaching and conveying strategies at a high standard and school personnel are delivery strategies at a high level.
Playground Intervention: Coach Ratings of Aide Implementation | Change from Exit to Follow Up (3 months follow up) in Playground Intervention Coach Rated Aide Fidelity
  Playground Intervention: Coach Rated Aide Fidelity. Fidelity forms will measure implementation mastery of interventionists and school personnel. This is to ensure that interventionists are teaching and conveying strategies at a high standard and school personnel are delivery strategies at a high level.
Playground Intervention: Observer Ratings of Aide Implementation | Change from baseline to exit (12 weeks later)
  Playground Intervention: Observer Rated Aide Fidelity. Fidelity forms will measure implementation mastery of interventionists and school personnel. This is to ensure that interventionists are teaching and conveying strategies at a high standard and school personnel are delivery strategies at a high level.
Playground Intervention: Observer Ratings of Aides Implementation | Change from exit to follow up (3 months later)
  Playground Intervention: Observer Rated Aide fidelity. Fidelity forms will measure implementation mastery of interventionists and school personnel. This is to ensure that interventionists are teaching and conveying strategies at a high standard and school personnel are delivery strategies at a high level.
STAT Intervention: Coach Rated Teacher Implementation | Change from baseline to exit (6 weeks)
  STAT Intervention: Coach Rated Teacher Fidelity. Fidelity forms will measure implementation mastery of interventionists and school personnel. This is to ensure that interventionists are teaching and conveying strategies at a high standard and school personnel are delivery strategies at a high level.
STAT Intervention: Coach Rated Teacher Implementation | Change from exit to follow up (3 months)
  STAT Intervention: Coach Rated Teacher Fidelity. Fidelity forms will measure implementation mastery of interventionists and school personnel. This is to ensure that interventionists are teaching and conveying strategies at a high standard and school personnel are delivery strategies at a high level.
STAT Intervention: Teacher Ratings of Implementation | Exit (12 weeks from Baseline)
  Climate for Implementation Measure is a 17-item questionnaire to measure the climate of each classroom. The survey asks teachers and aides to rate their perception of program quality and ease of use, and global perceptions of staff climate.
Playground Intervention: Aides Ratings of Effectiveness of Intervention | Change from Baseline to Exit (12 weeks later) in Playground Intervention Aide Rated Fidelity
  Playground Intervention Aide Rate Fidelity. Fidelity forms will measure implementation mastery of interventionists and school personnel. This is to ensure that interventionists are teaching and conveying strategies at a high standard and school personnel are delivery strategies at a high level.
STAT Intervention: Teachers Ratings of Effectiveness of Intervention | Change from Baseline to Exit (12 weeks later) in STAT Intervention in Teacher Fidelity
  STAT Intervention Teacher Fidelity. Fidelity forms will measure implementation mastery of interventionists and school personnel. This is to ensure that interventionists are teaching and conveying strategies at a high standard and school personnel are delivery strategies at a high level.
Playground Intervention: Aides Ratings of Effectiveness of Intervention | Change from Exit to Follow Up (3 months later) in Playground Intervention Aide Rated Fidelity
  Playground Intervention Aide Rated Fidelity. Fidelity forms will measure implementation mastery of interventionists and school personnel. This is to ensure that interventionists are teaching and conveying strategies at a high standard and school personnel are delivery strategies at a high level.
STAT Intervention: Teachers Ratings of Effectiveness of Intervention | Change from Exit to Follow up (3 months later) in STAT Intervention in Teacher Fidelity
  STAT Intervention Teacher's Fidelity. Fidelity forms will measure implementation mastery of interventionists and school personnel. This is to ensure that interventionists are teaching and conveying strategies at a high standard and school personnel are delivery strategies at a high level.

OTHER OUTCOMES:
Playground Intervention School Personnel Acceptability | Change from Baseline to Exit (12 weeks later) in Acceptability of Playground Intervention
  Playground Acceptability Scale is a 7-item questionnaire that uses a 5 point Likert Scale to rate acceptability
Playground Intervention: School Personnel Buy In of Intervention | Exit (12 weeks from baseline)
  The rate in which teachers and school personnel are accepting of the playground interventions strategies.
Playground Intervention: School Personnel Acceptability of Intervention | Change from Exit to Follow Up (3 months later) in Acceptability of Playground Intervention
  Playground Acceptability Scale is a 7-item questionnaire that uses a 5 point Likert Scale to assess acceptability of intervention.
STAT Intervention Teacher Buy In of Intervention | Exit (6 weeks from baseline)
  The rate in which teachers and school personnel are accepting of the STAT interventions.
Playground Intervention: Teacher's Social Opportunities Interview | At Baseline
  This interview captures the daily activities (and amount of time spent in those activities) of children with ASD in inclusive settings as well as the number of social opportunities children with ASD have with their peers throughout the school day (despite level of engagement in those activities).

CONTACTS AND LOCATIONS:
Overall Officials: Connie Kasari, Ph.D, Principal Investigator — University of California, Los Angeles; David Mandell, Sc.D, Principal Investigator — University of Pennsylvania; Tristram Smith, Ph.D, Principal Investigator — University of Rochester
Locations (3):
- United States (3):
  - UCLA Semel Institute, Los Angeles, California
  - University of Rochester Medical Center, Rochester, New York
  - UPENN Map Center for Mental Health Policy and Services Research, Philadelphia, Pennsylvania